CLINICAL TRIAL: NCT06159543
Title: The Effects of Fresh Mango Consumption on Cardiometabolic Outcomes in Free-living Individuals With Prediabetes: a Randomized Controlled Crossover Trial
Brief Title: The Effects of Fresh Mango Consumption on Cardiometabolic Outcomes in Free-living Individuals With Prediabetes
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Loma Linda University (Other)
Collaborators: National Mango Board (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 5230515
Record Dates: First submitted 2023-11-28; First posted 2023-12-06 (Actual); Last update posted 2025-10-06 (Actual); Status verified 2025-09

CONDITIONS: Hyperglycemia; Dyslipidemias; Insulin Resistance; Inflammation; Oxidative Stress
MeSH Terms: conditions — Hyperglycemia; Dyslipidemias; Insulin Resistance; Inflammation | interventions — Mangifera indica extract

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mango added to habitual diet (Experimental): Participants will be asked to consume 1.5 cups of mango per day for 12 weeks as part of their habitual diet.
  Interventions: Behavioral: Mango
- Habitual diet without mango (No Intervention): Participants will be asked to refrain consuming mangos for 12 weeks while continuing their habitual diet.

INTERVENTIONS:
Behavioral: Mango — 1.5 cups/day of mango for 12 weeks
  Arms: Mango added to habitual diet

SUMMARY:
The goal of this clinical trial is to test the effect of 12 weeks of 1.5 cups per day of fresh mango on glucose control, insulin resistance, lipids, inflammation, oxidation and body composition in individuals with prediabetes. The main questions it aims to answer are:

* What is the effect of 1.5 cups per day of fresh mango over 12 weeks on indicators of glycemic control including fasting glucose and HgbA1c?
* What is the effect of 1.5 cups per day of fresh mango over 12 weeks on fasting blood insulin and insulin resistance (HOMA-IR)?
* What is the effect of 1.5 cups per day of fresh mango over 12 weeks on lipids including LDL-cholesterol, total cholesterol, HDL-cholesterol and triglycerides?
* What is the effect of 1.5 cups per day of fresh mango over 12 weeks on oxidative stress including oxidized LDL-cholesterol and 8-iso-PGF2-alpha?
* What is the effect of 1.5 cups per day of fresh mango over 12 weeks on markers of inflammation including c-reactive protein, e-selectin, ICAM, VCAM, TNF-alpha and IL-beta?
* What is the effect of 1.5 cups per day of fresh mango over 12 weeks on percent body fat, fat mass, and lean mass?

Participants will be asked to:

* Consume 1.5 cups of mango per day for 12 weeks, take a 4 to 8 week break, and then avoid consuming mangos for 12 weeks
* Attend a prerandomization clinic prior to study
* Attend three (3) clinics where blood will be drawn during weeks 0, and 12 of the first phase and last week of the second phase of the study
* Attend eight (8) clinics where anthropometric measurements (height, weight, body composition) will be conducted and interaction with study clinicians will occur during weeks 0, 4, 8, 12 of each phase of the study
* Complete questionnaires and surveys in person and remotely, including six (6) 24-hour dietary recalls.

Researchers will compare the 12 weeks participants consume mango to the 12 weeks the participants are not consuming mango to see if there are differences in glycemic indicators, insulin resistance, lipids, inflammation, oxidation and body composition between the two time periods.

ELIGIBILITY:
Inclusion Criteria:

* HgbA1c of 5.7 to 6.4% indicative of prediabetes
* Abdominal obesity as defined as a waist circumference >102 cm for men or >88 cm for women

Exclusion Criteria:

* Self-reported chronic disease history (diabetes, heart disease, cancer, kidney disease, inflammatory bowel disease, etc.)
* Pacemaker
* Mango allergies
* Latex allergies (cross-reactive with mango)
* Smoking, use of tobacco, or high alcohol intake (>2 drinks/day for men or >1 drink per day for women)
* Recent significant weight loss (>5% within 6 months of study enrollment)
* BMI >35 kg/m^2
* Pregnancy or lactation
* Use of medication and/or supplements affecting glycemic indicators or lipids
* Habitual mango intake of >3 servings per week and/or habitual fruit intake of >2 servings per day
* Not able to read and/or communicate in English

Ages: 40 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 31 (Estimated)
Dates: Start 2024-07-30 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
LDL-cholesterol | LDL-cholesterol will be measured in fasting blood that will be drawn at weeks 0 and 12 of the first phase and the last week of the second phase of the study.
Total cholesterol | Total cholesterol will be measured in fasting blood that will be drawn at weeks 0 and 12 of the first phase and the last week of the second phase of the study.
HDL-cholesterol | HDL-cholesterol will be measured in fasting blood that will be drawn at weeks 0 and 12 of the first phase and the last week of the second phase of the study.
Triglycerides | Triglycerides will be measured in fasting blood that will be drawn at weeks 0 and 12 of the first phase and the last week of the second phase of the study.
HgbA1c | HgbA1c will be measured in fasting blood that will be drawn at weeks 0 and 12 of the first phase and the last week of the second phase of the study.
Fasting blood glucose | Fasting blood glucose will be measured in fasting blood that will be drawn at weeks 0 and 12 of the first phase and the last week of the second phase of the study.
Fasting blood insulin | Fasting blood insulin will be measured in fasting blood that will be drawn at weeks 0 and 12 of the first phase and the last week of the second phase of the study.
HOMA-IR (Insulin resistance) | Fasting blood glucose and insulin will be measured in fasting blood that will be drawn at weeks 0 and 12 of the first phase and the last week of the second phase of the study.
  Fasting blood glucose and fasting blood insulin will be used to quantify HOMA-IR values.
Oxidized LDL-cholesterol | Oxidized LDL-cholesterol will be measured in fasting blood that will be drawn at weeks 0 and 12 of the first phase and the last week of the second phase of the study.
8-iso-PGF2 alpha | 8-iso-PGF2 alpha will be measured in fasting blood that will be drawn at weeks 0 and 12 of the first phase and the last week of the second phase of the study.

SECONDARY OUTCOMES:
C-reactive protein | C-reactive protein will be measured in fasting blood that will be drawn at weeks 0 and 12 of the first phase and the last week of the second phase of the study.
E-selectin | E-selectin will be measured in fasting blood that will be drawn at weeks 0 and 12 of the first phase and the last week of the second phase of the study.
ICAM | ICAM will be measured in fasting blood that will be drawn at weeks 0 and 12 of the first phase and the last week of the second phase of the study.
VCAM | VCAM will be measured in fasting blood that will be drawn at weeks 0 and 12 of the first phase and the last week of the second phase of the study.
TNF-alpha | TNF-alpha will be measured in fasting blood that will be drawn at weeks 0 and 12 of the first phase and the last week of the second phase of the study.
IL-beta | IL-beta will be measured in fasting blood that will be drawn at weeks 0 and 12 of the first phase and the last week of the second phase of the study.
Percent body fat | Percent body fat will be measured at weeks 0, 4, 8, 12 of each phase of the study.
Fat mass | Fat mass will be measured at weeks 0, 4, 8, 12 of each phase of the study.
Lean body mass | Lean body mass will be measured at weeks 0, 4, 8, 12 of each phase of the study.

CONTACTS AND LOCATIONS:
Overall Officials: Celine Heskey, DrPH, Principal Investigator — Loma Linda University
Locations (1):
- Nutrition Research Center, School of Public Health, Loma Linda University, Loma Linda, California, United States